CLINICAL TRIAL: NCT01546376
Title: Observational Study of Effect of Radiation Therapy to Immuno Status in HIV-cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: THAIHIV001
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2009-01

CONDITIONS: To Study Immunostatus of HIV-cancer Patients Who Recived RT Befor RT and Last Week of RT; To Study HIV Viral Load of HIV-cancer Patients Who Recived RT Befor RT and Last Week of RT
MeSH Terms: interventions — Radiotherapy; Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-cancer patients who recived RT
  Interventions: Radiation: Radiation therapy; Other: Venepuncture

INTERVENTIONS:
Radiation: Radiation therapy — External photon beam radiation therapy dosage 4000-7000 CGy
Other: Venepuncture — Venepuncture for CD4 and viral load count at Week 0, Last week of Radiation, and 12, 24 Week follow up

SUMMARY:
Objectives: To study immunostatus (CD4) and HIV viral load in HIV-cancer patients before RT and last weeks of RT .

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* HIV positive cancer patients
* Photon beam RT, conventional fraction >= 4000 cgy in 4 weeks

Exclusion Criteria:

* CD4 count < 200 cell/ml and not received anti retro viral

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV positive cancer patients Curative RT treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-08

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand